CLINICAL TRIAL: NCT06625294
Title: Comparative Effects of Constraint-Induced Movement Therapy With Bilateral Functional Task Training On Hand Function In Patients With Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/32
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Hand Function
Keywords: Task Oriented Training; Constraint-Induced Movement Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group A (Experimental): It includes participants receiving task oriented combined with bilateral functional task training exercises for 10 weeks treatment.
  Interventions: Procedure: Task -oriented training with bilateral functional task training exercises
- Experimental group B (Experimental): This group involves participants receiving task oriented training with constrained induced movement therapy exercises for a period of 10 weeks.
  Interventions: Procedure: Task Oriented Training with CIMT

INTERVENTIONS:
Procedure: Task -oriented training with bilateral functional task training exercises — Task oriented training approach with BFTT will consists of different tasks including:
  Hand Movements:
  1. Fold a small cloth towel with both hands with initially putting the towel flat on the table and gradually folding it into a large towel roll.
  2. Put a small amount of putty on patient's table and instruct to roll it with the help of rolling pin moving it back and forth using both the hands.
  3. Place a jar with a removable lid on the table and instruct the patient to remove lid from the jar completely by holding the jar with either hand and remove the lid with the alternate hand.
  4. Pouring water: Pour water from jug while holding the jug in unaffected hand to cup/glass that is held in affected hand and activity can be done the other way round as well.
  5. Pour water from one hard plastic cup to another while alternatively involving both the hands (we must not allow deformation of the cup)
  6. Plunging action with coffee maker against water resistance:Fill the coffee maker with water.
  Arms: Experimental group A
Procedure: Task Oriented Training with CIMT — • Hand Movements:
  1. Sitting at a table (Wrist Extension): Affected forearm resting on table. Place cylindrical object in palm of patient's hand. Patient asked to move the hand towards the forearm (dorsiflexion) by extending the wrist - no elbow flexion allowed.
  2. Sitting at a table (Radial Deviation of Wrist): Therapist should place forearm with ulnar side on table in mid-pronation / supination position. Thumb in line with forearm and wrist in extension. Fingers around cylindrical object. Patient is asked to lift hand off table. No wrist flexion or extension.
  Advanced Hand Activities:
  1. Have the patient reach forward to pick up the top of a pen with their affected hand, bring the affected arm back to their side and put the pen cap down in front of them.
  2. Place (beans), in a teacup an arm's length away on the affected side. Place another teacup an arm's length away on the intact side. Have the patient pick up one beans with their affected hand and place the beans in the cup on the
  Arms: Experimental group B

SUMMARY:
Task-oriented training is an approach that will encourage active participation of the patient making treatment functional and task orientated in order to achieve the best possible recovery following injury.

Neurorehabilitation studies have shown that Constrained induced movement therapy can increase both motor function and the use of the paretic arm and that these improvements parallel changes in the activation of the brain sensorimotor network.

Bilateral Functional Task Training which promotes the use of the paretic limb simultaneously with the nonparetic limb. Many of our daily chores are bimanual and utilize concurrent use of both arms.

DETAILED DESCRIPTION:
OBJECTIVES:

The objectives of this study are:

1. To determine the effects of constraint induced movement therapy post-stroke patients with motor impairment of hand in terms of grasp/grip, pinch and gross movements.
2. To determine the effects of bilateral functional task training post-stroke patients with motor impairment of hand in terms of grasp/grip, pinch and gross movements.
3. To determine the comparative effects of constraint, induced movement therapy versus bilateral functional task training post-stroke patients with motor impairment of hand in terms of grasp/grip, pinch and gross movements.

HYPOTHESIS:

Alternate Hypothesis:

1. There will be significant effect of constraint induce movement therapy versus bilateral functional task training on hand function in patients with stroke in terms of grasp/grip p<0.05
2. There will be significant effect of constraint induce movement therapy versus bilateral functional task training on hand function in patients with stroke in terms of pinch and gross movements. p<0.05

Null Hypothesis:

1. There will be no significant effect of constraint induce movement therapy versus bilateral functional task training on hand function in patients with stroke in terms of grasp/grip p<0.05
2. There will be no significant effect of constraint induce movement therapy versus bilateral functional task training on hand function in patients with stroke in terms of pinch and gross movements. p<0.05

Research Design: Experimental study. Randomized Control Trial

Clinical setting: Neuromedicine Department,Neurology OPD,Rehab OPD, Multidisciplinary Lab in FUCP, Fauji Foundation Hospital and Treatment room FUCP.

Study duration: 1 year

Selection Criteria:

Inclusion Criteria

1. Both genders.
2. Age range from 40 to 60years.
3. Diagnosed Cases of Stroke.
4. MMT greater than Grade 2.
5. Wrist ROM valid for functional tasks.
6. Brunnstrom stages of recovery: Grade 4
7. MAS: Grade 2 or less

Exclusion Criteria

1. Active joint disease (rheumatoid, or any other rheumatological disease)
2. Recent history of upper limb surgery.
3. Contractures or Deformity.
4. Inability to follow-2-step commands.
5. Psychiatric diagnoses.

Technique: Convenience Sampling

Outcome Measures:

Data will be collected on Demographics and general information. Data will be collected using Action research arm test,Fugl-Meyer Assessment Upper Extremity (FMA-UE),Goniometry.

Experimental Group (A) = This group will receive task oriented training with bilateral functional task training and their outcomes will be measured at baseline and at the end of 10 weeks treatment..

Control group (B) =This group will undergo task oriented training with Constrained Induced Movement Therapy and their outcomes will be observed at the baseline and then after treatment of 10 weeks.

Data analysis techniques:

The data will be analyzed through SPSS 21 and Data would be analyzed based on the study design chosen that is random control experimental study within the community.

A printed questionnaire will be provided to the patients after obtaining written consent and providing adequate explanation regarding the study, after which the data will be presented in the form of graphs or tables.

Significance of the study:

1. Task oriented training program including Constraint Induced movement therapy and Bilateral Functional Task Training for the restoration and improvement of the hand function in patients with stroke will prove effective in increasing strength and improving function along with grasp /grip pinch and gross movements.
2. This study will help the practitioner to use the new treatment comparison options for treating patient's hand function improvement in stroke.
3. The results of the study will add to the literature about the comparative effects of Constraint Induced movement therapy and Bilateral Functional Task Training in improving hand function in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age range from 40 to 60 years.
* Diagnosed Cases of Stroke.
* MMT greater than Grade 2.
* Wrist ROM valid for functional tasks.
* Brunnstrom stages of recovery: Grade 4
* MAS: Grade 2 or less Exclusion Criteria
* Active joint disease (rheumatoid, or any other rheumatological disease)
* Recent history of upper limb surgery.
* Contractures or Deformity.
* Inability to follow-2-step commands.
* Psychiatric diagnoses.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Upper extremity performance | 10 weeks
  Action Research Arm Test (ARAT) will be used for estimation of upper-limb function. This is a summated rating scale with 4 domains: Grasp, Grip, Pinch, and Gross. Scoring is based on the performance of several tasks from each domain. Each task is rated from 0 to 3, where higher scores denote less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Zahid, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan